CLINICAL TRIAL: NCT00126100
Title: A Randomized Clinical Trial of Stem Cell Mobilization by Granulocyte-Colony-Stimulating Factor in Patients With Acute Myocardial Infarction. Regenerate Vital Myocardium by Vigorous Activation of Bone Marrow Stem Cells (REVIVAL-2) Trial
Brief Title: Bone Marrow Stem Cell Mobilisation Therapy for Acute Myocardial Infarction (AMI)(REVIVAL-2)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Wilhelm Sander Foundation (Unknown); Schulz Foundation (Unknown); Else Kröner Fresenius Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. I01003; KKF 10-02; KKF 04-03
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Myocardial Infarction
Keywords: Stem Cells
MeSH Terms: conditions — Myocardial Infarction | interventions — Filgrastim; Lenograstim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients were randomly assigned to receive subcutaneously a daily dose of 10 microg/kg of G-CSF for 5 days.
  Interventions: Drug: G-CSF Granulocyte-Colony Stimulating Factor
- 2 (Placebo Comparator): Patients were randomly assigned to receive subcutaneously a daily dose of placebo for 5 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: G-CSF Granulocyte-Colony Stimulating Factor — Patients were randomly assigned to receive subcutaneously a daily dose of 10 microg/kg of G-CSF for 5 days.
  Other Names: Neupogen (Filograstim); Granocyte (Lenograstim)
  Arms: 1
Other: Placebo — Patients were randomly assigned to receive subcutaneously either a daily dose of 10 microg/kg of G-CSF or placebo for 5 days.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether stem cell mobilization by granulocyte colony-stimulating factor (G-CSF) therapy in patients with acute myocardial infarction after successful mechanical reperfusion reduces infarct size.

DETAILED DESCRIPTION:
Experimental studies and early-phase clinical trials suggest that transplantation of blood-derived or bone marrow-derived progenitor cells may improve cardiac regeneration after acute myocardial infarction. Granulocyte colony-stimulating factor (G-CSF) induces mobilization of bone marrow stem cells and, thereby, increases the number of circulating stem cells that are available cells for myocardial regeneration.

ELIGIBILITY:
Inclusion Criteria:

* ST-elevation acute myocardial infarction (5 days before randomization)
* Successful percutaneous coronary intervention [PCI] (performed within 12 hours from symptom onset)
* Scintigraphic infarct size >5% of left ventricle
* Written informed consent

Exclusion Criteria:

* Age <18 years or >80 years
* Congestive heart failure defined as Killip class >2
* A history of myocardial infarction
* Electrical or hemodynamic instability
* Autoimmune diseases
* Fructose intolerance
* Malignancies
* Incompatibility of filgrastim
* Known or suspected pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2004-02; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Reduction of infarct size (measured by Tc-sestamibi scintigraphy) | measured by Tc-sestamibi scintigraphy baseline, 4 and 6 months

SECONDARY OUTCOMES:
Left ventricular ejection fraction | Left ventricular ejection fraction
Incidence of angiographic restenosis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schomig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum, Munich
  - 671. Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Orlic D, Kajstura J, Chimenti S, Limana F, Jakoniuk I, Quaini F, Nadal-Ginard B, Bodine DM, Leri A, Anversa P. Mobilized bone marrow cells repair the infarcted heart, improving function and survival. Proc Natl Acad Sci U S A. 2001 Aug 28;98(18):10344-9. doi: 10.1073/pnas.181177898. Epub 2001 Aug 14. PMID 11504914
- [Background] Kocher AA, Schuster MD, Szabolcs MJ, Takuma S, Burkhoff D, Wang J, Homma S, Edwards NM, Itescu S. Neovascularization of ischemic myocardium by human bone-marrow-derived angioblasts prevents cardiomyocyte apoptosis, reduces remodeling and improves cardiac function. Nat Med. 2001 Apr;7(4):430-6. doi: 10.1038/86498. PMID 11283669
- [Background] Harada M, Qin Y, Takano H, Minamino T, Zou Y, Toko H, Ohtsuka M, Matsuura K, Sano M, Nishi J, Iwanaga K, Akazawa H, Kunieda T, Zhu W, Hasegawa H, Kunisada K, Nagai T, Nakaya H, Yamauchi-Takihara K, Komuro I. G-CSF prevents cardiac remodeling after myocardial infarction by activating the Jak-Stat pathway in cardiomyocytes. Nat Med. 2005 Mar;11(3):305-11. doi: 10.1038/nm1199. Epub 2005 Feb 20. PMID 15723072
- [Result] Zohlnhofer D, Ott I, Mehilli J, Schomig K, Michalk F, Ibrahim T, Meisetschlager G, von Wedel J, Bollwein H, Seyfarth M, Dirschinger J, Schmitt C, Schwaiger M, Kastrati A, Schomig A; REVIVAL-2 Investigators. Stem cell mobilization by granulocyte colony-stimulating factor in patients with acute myocardial infarction: a randomized controlled trial. JAMA. 2006 Mar 1;295(9):1003-10. doi: 10.1001/jama.295.9.1003. PMID 16507801